CLINICAL TRIAL: NCT02676999
Title: Clinical and Radiographical Analysis of the Distal Radioulnar Joint Following Implantation of a Scheker Total Distal Radioulnar Joint Prosthesis
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0369
Record Dates: First submitted 2015-01-14; First posted 2016-02-09 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2016-02

CONDITIONS: Scheker Total Distal Radioulnar Joint Prosthesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months

INTERVENTIONS:
Procedure: Implantation of a Scheker total distal radioulnar joint prosthesis

SUMMARY:
This project is set to describe by objective measures as the range of motion and weight-bearing ability of the distal radioulnar joint one to five years after primary implantation of a Scheker total distal radioulnar joint prosthesis.The range of motion and stability of the distal radioulnar joint (DRUJ) are important outcomes to preserve function, especially the pronation and supination. Unlike other ulnar endoprostheses that replace only the ulnar head, the Scheker prosthesis replaces the ulnar head, resurfaces the lesser sigmoid notch, and is semi-constrained in design.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with a Scheker total distal radioulnar joint prosthesis and with a follow-up time between 12 and 60 months after primary implantation
* Patient willing and able to give written informed consent to participate in the study

Exclusion criteria:

* Inflammatory disease (e.g. rheumatoid arthritis)
* Pregnant women
* German language barrier to complete the questionnaires
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Legal incompetence
* Participation in any other medical device or medicinal product study within the previous months that could influence the results of the present study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient treated with a Scheker total distal radioulnar joint prosthesis and with a follow-up time between 12 and 60 months after primary implantation, who were willing and able to give written informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Primary outcomes of this study are active DRUJ range of motion (pronation and supination) and weight-bearing ability in neutral and pronated position. | Follow-up time between 12-60 months after primary implantation of the Scheker prothesis

SECONDARY OUTCOMES:
Secondary outcomes of this study are radiological parameters, pain level by Visual Analog Scale, objective functional parameters (passive stability, grip strength), subjective functional parameters, and complications affecting the examined wrist. | Follow- up time between 12-60 months after primary implantation of the Scheker prothesis

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Center for Reconstructive Surgery, Zurich, Canton of Zurich, Switzerland